CLINICAL TRIAL: NCT04020705
Title: The Efficacy of Citicoline in Eyedrops (OMK1) in Reducing the Progression of Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto di Ricerca Neuroftalmologia S.r.l. (Network)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Luca Rossetti, Director Clinical Ophthalmologist P.O. San Paolo Milan, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMK20115
Record Dates: First submitted 2019-04-12; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Glaucoma
Keywords: Glaucoma; Glaucoma Open Angle; Pseudoexfoliation Glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Exfoliation Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citicoline eye drops (OMK1) (Experimental): 45 patients will be treated with active treatment (OMK1)
  Interventions: Device: Citicoline eye drops (OMK1)
- hypromellose based ocular lubricant (Placebo Comparator): 45 patients will be treated with placebo (lubricant eye drops)
  Interventions: Other: Placebo Comparator: hypromellose based ocular lubricant

INTERVENTIONS:
Device: Citicoline eye drops (OMK1) — (OMK1) will be prescribed in the dosage of 1 drop 3 times a day
  Arms: Citicoline eye drops (OMK1)
Other: Placebo Comparator: hypromellose based ocular lubricant — will be prescribed in the dosage of 1 drop 3 times a day
  Arms: hypromellose based ocular lubricant

SUMMARY:
Double-blind study (OMK1 vs. Placebo) A total of 90 patients, 30 per center, will be the study sample. The study will include patients with Primary Open angle Glaucoma (glaucoma or pseudoexfoliation) with a loss of visual field with MD between -2 dB and -15 decibel.

Patients will be randomized into 2 treatment groups, both treated with hypotonic ocular drug therapy: one part of the patients will be treated with the OMK1 Medical Device containing topical citicoline for 3 years; the remaining part will receive a placebo.

All patients will be followed with quarterly visits which will check, in addition to the intraocular pressure (IOP), the structure of the optic nerve and visual function (standard visual field).

The primary objective is to evaluate a reduction of the perimetric progression in the group that receives the topical citicoline compared to the group treated with placebo. The reduction of the progression will be evaluated with Spectral Domain Optic coherence tomography and with standard perimetry (SAP).

The secondary objective is to assess the tolerability and safety of OMK1 eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Patients with POAG and pseudoexfoliation glaucoma in one or both eyes. In the latter case, only one eye (chosen at random) will be used for the analysis.
* Patients with -2 < MD < -15 dB, progression of MD at least -0,5 dB/y for 2 years.
* Patients with tonometric compensation, i.e., IOP not above 18 mmHg. Tonometric compensation can be achieved with any type of hypotonic medical therapy and must be maintained during the 3 years of the study. If at any check-up the average of at least 3 measurements of IOP at different times is higher than 18 mmHg, the patient will be offered a new hypotonic treatment (including surgery) to control the progression of the disease. If compensation cannot be achieved (e.g., the patient refuses the proposed therapy or, in spite of this does not achieve satisfactory IOP values), the patient will be excluded from the study.
* Patients over the age of 18 years

Exclusion Criteria:

* Patients with contraindications to citicoline
* Patients with IOP higher than 18 mmHg
* Patients with other forms of glaucoma
* Patients treated with other neuroprotective therapies
* Women who are pregnant and/or breastfeeding
* Pediatric or adolescent patients aged under 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Change in glaucomatous damage | Baseline and Visit at 36 months
  The primary objective of the study is to assess whether there is a difference in the deterioration of glaucomatous damage with standard perimetry (HFA 24-2 and 10-2) in the group that receives the topical citicoline in addition to topical therapy with hypotensive drugs compared to the group treated with the sole reduction of intraocular pressure.

SECONDARY OUTCOMES:
progression of glaucoma in the SD OCT examination | Baseline and Visit at 36 months
  assessment of the progression of glaucoma in the SD OCT examination (Retinal Nerve fiber Layer- RNFL evaluation) in the group that receives the topical citicoline together with ocular antihypertensive drug therapy compared to the group treated with the sole reduction of intraocular pressure.
  It will be used for the assessment of the progression of glaucoma the Brusini staging system.

IPD SHARING:
Plan to Share IPD: No